CLINICAL TRIAL: NCT00869076
Title: Pharmacist Management of Diabetes Mellitus: A Randomized Controlled Trial.
Brief Title: Pharmacists Management of Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advantage Health Physician Network (Other)
Collaborators: Doran Foundation (Unknown); Michigan Pharmacist Foundation (Unknown); Priority Health (Unknown); Western Michigan Society of Health System Pharmacists (Unknown)
Responsible Party: John Jameson, PharmD., Ferris State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PharmacistDiabetesJameson
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Pharmacist
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist Management (Experimental): In this arm the Pharmacist managed the Diabetes in collaboration with the primary care physician
  Interventions: Other: Pharmacist Management
- Usual Care (Active Comparator): The patient was managed by the primary care physician
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pharmacist Management — Pharmacist Managed the patient's diabetes in collaboration with their primary care physician
  Arms: Pharmacist Management
Other: Usual care — Patient was managed by their primary care physician as usual
  Arms: Usual Care

SUMMARY:
The hypothesis is that patients with poorly controlled diabetes would have greater improvement in their blood sugar control when managed by a clinical pharmacist than when managed with usual medical care. Patients with poor control are randomized to pharmacist management or to usual medical care for one year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* A1c greater than or equal to 9.0

Exclusion Criteria:

* Not expected to live for the duration of the study
* Managed by an endocrinologist
* Unwillingness to participate and attend pharmacist visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Hgb A1c change | 1 year

SECONDARY OUTCOMES:
HgbA1c change based on ethnicity | one year
percent of patients with a 1 point or greater decrease in A1c | one year
Percent of patients with a 1 point decrease in A1c by ethnicity | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Advantage Health Physican Network, Grand Rapids, Michigan, United States